CLINICAL TRIAL: NCT05642169
Title: Effect of a High Interval Intensity Training Program on Quality of Life, Mental Health, Brain Executive Functions, and IGF-1 Response in Sedentary Young University Women.
Brief Title: Effect of a HIIT Program on Quality of Life, Executive Functions, and IGF-1 Response in Sedentary Young University Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Jimenez-Roldan Manuel Jesus, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Young Brain Proyect
Record Dates: First submitted 2022-11-18; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Insulin Growth Factor I Deficiency; IGF1 Deficiency; Executive Function Disorder
Keywords: HIIT; IGF-1; young adult; women
MeSH Terms: conditions — Insulin-Like Growth Factor I Deficiency

STUDY DESIGN:
Intervention Model Description: The present research follows a randomized controlled experimental design (RCT), sequential type, with parallel groups with three groups and repeated measures, being evaluated in a pretest, posttest and after the end of the follow-up period.
  The sample, of casual or incidental type, were randomly distributed in two experimental groups and one CG, thus avoiding selection bias. The CG continued to maintain their lifestyle on a daily basis. On the other hand, we found two experimental groups, which performed a HIIT program with a frequency of 3 workouts per week. In one of them (HIIT+AF), the focus was on increasing their daily physical activity through the execution of 10,000 steps per day. The other experimental group (HIIT) followed the same HIIT program.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT (Experimental): Training program for 12 weeks with a frequency of 3 workouts per week.
  Interventions: Behavioral: HIIT
- HIIT+AF (Experimental): They will develop the same training program as the HIIT group, and they will also have to perform 10,000 steps per day.
  Interventions: Behavioral: HIIT+PA
- Control (Placebo Comparator): They will not suffer any change in their lifestyle.
  Interventions: Behavioral: CON

INTERVENTIONS:
Behavioral: HIIT — The training sessions will have a frequency of 3 times per week (Monday, Wednesday and Friday) and the duration will be between 39 to 54 minutes, depending on the training week.
  The training program will be developed with the own body weight of each participant. Therefore, a progression according to the needs of this population will be fulfilled. The session model could be multi-joint exercises with self-loads, where the difficulty of the exercises will be worked progressively. Throughout the main part of each workout, 30 seconds of work will be performed at the corresponding intensity and 30 seconds of rest. Halfway through the total repetitions, there will be 2 minutes of recovery.
  Arms: HIIT
Behavioral: HIIT+PA — In relation to the 2 groups that will perform HIIT, the HIIT+AF will have to complete 10.000 steps per day. In this way, they will be focusing on increasing their daily physical activity. In addition, this group will perform the same HIIT training programme as the other experimental group.
  Arms: HIIT+AF
Behavioral: CON — This group will not suffer any changes in their lifestyle
  Arms: Control

SUMMARY:
Sedentary lifestyle, understood as an activity that requires minimal body movement (Tremblay et al., 2017), is one of the main factors responsible for chronic diseases in Young adults.

In addition, this sedentary lifestyle generates mental disorders, such as anxiety, low self-esteem and depression, being more pronounced in women than in men (Nihill et al., 2013). Thus, both daily physical activity (PA) and physical exercise programs (PE), of moderate-vigorous intensity, act as an effective tools for the improvement of quality of life, since they generate benefits at physiological, psychological and social levels (Cohen et al., 2019).

If we focus on young adult, it can be seen how there is a significant decrease in the practice of physical exercise at this age (Grim et al., 2011). This means that the aforementioned recommendations are not reached (Cancela et al., 2019). Furthermore, if compared between sexes, lower levels are shown in the female sex (King et al., 2014).

For this reasons, and taking into account that the female population is a population vulnerable to significantly reduce their physical activity practice with age (Cohen et al., 2019), it is interesting to investigate on the possible health-related factors that this entails, such as quality of life, physical condition and mental health.

For these reasons, it is necessary to create effective strategies to address factors related to the main cognitive impairments and thus preserve better mental health.

Among all possible strategies, both pharmacological and non-pharmacological for the improvement of mental health, cognition and executive functions in young adults.Physical exercise has been shown to be a highly effective strategy at these ages (Heath et al., 2016). The stimulation of HIIT seems to reduce antioxidant responses. In recent years, there is a high interest in knowing the effect of HIIT on different health outcomes, such as physical and psychological fitness (Eather et al., 2019).

For all these reasons, sedentary lifestyles are an important public health factor associated with numerous pathologies and have been shown to have a significant cognitive involvement. Although we know that physical exercise can have a preventive role in the management of these associations, the conditioning factors of physical exercise are unknown, as well as the lifestyle factors that could contribute to a greater extent to the improvement of executive functionality in young women.

DETAILED DESCRIPTION:
The present investigation follows a randomized controlled experimental design (RCT), of sequential type, with parallel groups with three groups and repeated measures, being evaluated in a pretest, posttest and after the end of the follow-up period.

The sample, of casual or incidental type, was randomly distributed in two experimental groups and a control group, thus avoiding selection bias.

Once the study population had been selected and met the established inclusion and exclusion criteria, a 12-week HIIT-based intervention was performed.

Two of the experimental groups will perform this training program with the only difference that the HIIT+PA group will have to perform 10,000 steps per day, thus increasing daily physical activity.

Among the main study variables were insulin-like growth factor-1 (IGF-1), executive functions, physical condition, physical activity, quality of life and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-30 years old
* Reflect in the IPAQ questionnaire to be in category 1 or low level of physical activity (Craig et al., 2003) and therefore not conform to the minimum recommendations for physical activity and physical exercise proposed by the WHO.
* Not suffering from somatic signs or serious psychiatric illnesses that prevent the practice of physical exercise.
* Not attending psychological therapies in the last 12 months prior to the study. The use of this type of treatment may have an impact on the improvement of cognitive abilities and executive functions of the study population.
* Being able to communicate.
* Informed consent: Be able and willing to give informed consent.

Exclusion Criteria:

* Having a general cognitive impairment or executive function disorder recognized and treated by specialists.
* Physical activity: In order to select sedentary subjects, we excluded those who engaged in physical activity in their leisure time in a continuous and planned manner.
* Bilingualism: Habitual and indistinct use of two or more languages. This may condition the results in various cognitive tests present in the study, since it is known that this intellectual capacity has a morphological and functional impact on the brain.
* Musical instrument: Playing a musical instrument regularly and continuously, as in the previous criterion, generates a positive effect on the subject's cognition

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — There are gender differences in the practice of physical activity, being lower in women than in men in young adults. This leads to changes in different aspects, such as quality of life, physical and mental health. Among the state of mental health, differences have been observed in executive functions between men and women, sometimes being more reduced in the latter.
Enrollment: 75 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Biochemical determinants | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  The main biochemical determinants established in this study will be measured in saliva. Thus, the magnitude of the IGF-1 response in saliva as a consequence of the execution of a 12-week HIIT training program will be analyzed. In addition, the acute response to maximal effort will be measured at the initial and final assessments.
  Saliva will be collected in a fasted state (between 8-12 hours) and the passive drooling method will be used. At each assessment, a saliva sample will be obtained at rest and after maximal effort.
  To measure the variability in each assessment of IGF-1 concentration in saliva, the ELISA KIT protocol will be used.

SECONDARY OUTCOMES:
Body composition | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  Body composition will be measured by taking waist and hip perimeters and through electrical bioimpedance (BIA). This is a fast and non-invasive technique in which different body composition variables are estimated. Such a tool becomes a reliable system with scientific validity (Kelly & Metcalfe, 2012).
  The BIA used in this investigation (Tanita BC-418, Tokyo, Japan) is a segmental measurement. The subject is placed in a standing position on 4 electrodes, located on the feet and hands, where through two of them an alternating current is introduced and the remaining two collect this current, measuring, among others, the values of impedance, resistance and body reactance.
Maximum oxygen consumption | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  Maximum oxygen consumption (VO2max) will be estimated from the maximum power output (MPO) achieved in an incremental cycloergometer test (Andersen, 1995). Therefore, only the MPO will be taken into account for its estimation, since it is a measure of the capacity of the cardiorespiratory system, which can predict 80% of the variation in VO2max.
  The development of the test begins with a first part of 7 minutes at a submaximal load of 69W. At the end of this phase the heart rate was recorded with a pulsometer (H10 Polar Electro OY, Finalandia). The load will be increased by 35W every 2 minutes until the subject reached exhaustion.
Physical activity and sedentary behaviour | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  Physical activity will be evaluated objectively by accelerometry. The accelerometer is a device that allows objective quantification of the physical activity performed by a person. The study population was asked to wear a triaxial accelerometer (GTX3, Penascola, Florida, USA).
  Participants were instructed to wear the accelerometer throughout the day (24h). The placement of the accelerometer during the recording days should be on the right side at hip height and in line with the anterior face of the ipsilateral lower extremity. To avoid damage to the device, it was removed in any aquatic situation. On this occasion, a record sheet was provided for its annotation.
SF-36 quality of life. | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  To detect changes in health-related quality of life, the SF-36 questionnaire will be used. This questionnaire, in its Spanish versión (Vilagut et al., 2005), focuses on assessing general health status through a generic scale. This provides a profile of quality of life, both of a general population and of specific subgroups.
  This questionnaire consists of a total of 36 questions covering 8 health concepts. In addition, there are two summary measures, which are physical health and mental health. Mental health is divided into the vitality scale (4 items), social functioning (2), emotional role (3) and mental health (5). On the other hand, physical health encompasses physical capacity (10 items), physical role (4), bodily pain (2) and general health (5). In addition, two global questions on the perception of their health are added.
  The scores for each scale range from 0 to 100, with higher scores indicating a better quality of life
Rosenberg self-esteem scale. | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  The Rosenberg self-esteem scale (1965) is the most widely used test for the evaluation of self-esteem in scientific research and clinical practice.
  This test is a 10-item scale for analyzing global self-esteem (Vázquez Morejón et al., 2004). Each item is classified on a 4-point Likert scale, where 1 is equivalent to "strongly disagree" and 4 to "strongly agree". Of the 10 questions asked, five are formulated positively and five negatively (2,5,8,9,10). In addition, each question measures the degree of satisfaction of the person together with the person's self-assessment.
  In relation to the results, the unifactorial nature proposed by Rosenberg has been questioned; however, other authors support a bifactorial structure of positive and negative self-esteem. According to the validation study of this work in Spanish (Atienza et al., 2000), when the sample is made up of women, the elaboration of a single factor of global self-esteem is suggested.
Hamilton Rating Scale for the Evaluation of Depression (HDRS). | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  The HDRS (Hamilton, 1960) is a scale for assessing depression. It is hetero-applicable and is designed with the aim of quantitatively assessing the degree of depression of the interviewed subject.
  The original version consists of 21 questions, but on this occasion the reduced versión (Hamilton, 1967) published later will be used. This version consists of 17 questions, which is recommended for clinical use.
  The short version of the HDRS has been validated in the Spanish version (Ramos-Brieva & Cordero Villafáfila, 1986) showing high reliability and sensitivity to change in different populations (Ramos-Brieva & Cordero-Villafafila, 1988).
Executive functions | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  The measurements of the following cognitive tests will be performed with the collaboration of a psychologist specialized in the execution and description of the following executive tests:
  For the evaluation of inhibitory control, the Stroop testT will be used (Golden, 1999). This is a neuropsychological test that measures the interference generated in the performance of a task. In this work, the Victoria version will be developed in a digitized form (Mueller et al., 2012).
  For the evaluation of cognitive flexibility, wil be used the Wisconsin card test (WCST) (Cepeda et al., 2000). It can be performed traditionally or, as in this case, digitally. This test consists of a total of 64 cards. The cards present different combinations according to 4 geometric shapes, 4 colors and 4 quantities.
  Digit Span Test (DST) analyzes the ability to store and retain information, whose mission is to measure working memory.
Lower body muscle strength | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  Leg extension muscle strength will be assessed on a calibrated isokinetic dynamometer (Biodex System 4, Biodex Medical System, Inc., Shirley, NY, USA). Therefore, the Biodex System 4 will be used to assess each subject's ability to generate maximal isometric power with the knee extensor musculature in a 60° flexion joint position from a seated position.
  For measurement, the Biodex clinical data station will be used to analyze the Biodex torque and position signals and obtain the resulting measurements.
  The performance protocol will consist of executing two maximal isometric efforts for 5 seconds. The subject, with arms crossed over the chest, will begin to perform the maximal force at the evaluator's "push" voice. Subsequently, the subject will rest 30 seconds to perform the second attempt.
  Once both attempts have been completed, the best result of the peak torque variable (N-M) will be recorded for further analysis.
Upper extremity muscle strength. | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  Upper extremity muscle strength will be assessed through manual dynamometry testing with a digital dynamometer (TKK 5101 Grip-D; Takey, Tokyo, Japan) as described in other studies (Ruiz-Ruiz et al., 2002).
  Subjects were to be placed in a bipedal position during the test with the arms in full extension and without touching any part of the body with the dynamometer, except for the hand. The positioning of the body should be at all times with the shoulder girdle parallel to the ground, without allowing flexion or lateral movement of the trunk during the application of force.
  The participants will be instructed to squeeze the dynamometer grip as hard as possible and without being able to bend any of the joints involved. The duration of the effort will be 5 seconds, without being able to perform discontinuous activations, i.e., they must maintain the maximum isometric force possible during the 5 seconds.
  Finally, the best result (Kg) of the two tests performed will be recorded.
Beck Depression Inventory (BDI-II) | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  The Beck-II (Beck & Steer, 1993) is used to measure depressive symptomatology.
  It is a self-administered instrument consisting of 21 items that assess cognitive, affective and neurovegetative factors. This questionnaire is usually the most widely used in clinical psychology to assess the degree of depression (Sanz et al., 2003).
  This questionnaire has been validated in the Spanish version (Sanz et al., 2005) and has also shown high reliability in a university population (Sprinkle et al., 2002).
  Each item has four responses, ordered from least to most severe (from 0 to 3 points), and the subject must choose the sentence that most closely matches his or her perception during the last week. The scores of this instrument range from 0-63, with the reference cut-off points being the following: 0-9 no depression; 10-15 mild depression; 16-19 moderate depression; 20-29 moderate-severe depression; 30-63 severe depression.
International Physical Activity Questionnaire (IPAQ). | Up to 12 weeks (post) and through study completion, an average of 24 weeks (Follow-Up).
  The IPAQ questionnaire is an instrument to determine approximately the level of physical activity practiced by the general population (Hagstro et al., 2006). This questionnaire is one of the most widely used for the detection of sedentary lifestyles, used to a greater extent in its short version, adapted and translated into Spanish. In addition, this questionnaire shows excellent reliability (Craig et al., 2003) and high validity for its application in university population (Cancela et al., 2019).
  Therefore, for the calculation of the IPAQ data, an average of Mets will be adopted for each type of activity, resulting as follows: walking 3.3 Mets, moderate activities 4.0 Mets and intense activities 8.0 Mets.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Jesus Jimenez Roldan, Principal Investigator — University of Seville
Locations (1):
- Education Faculty, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang Y, Zhang B, Gan L, Ke L, Fu Y, Di Q, Ma X. Effects of Online Bodyweight High-Intensity Interval Training Intervention and Health Education on the Mental Health and Cognition of Sedentary Young Females. Int J Environ Res Public Health. 2021 Jan 3;18(1):302. doi: 10.3390/ijerph18010302. PMID 33401605
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33401605/